CLINICAL TRIAL: NCT01518582
Title: The GRANVIA®-C Cervical Disc Prosthesis to Treat Symptomatic Degenerative Disc Diseases
Brief Title: GRANVIA®-C Cervical Disc Prosthesis Multicenter European Pilot Study
Status: Completed | Type: Observational
Sponsor: Medicrea International (Industry)
Responsible Party: Sponsor
Other Study IDs: #0802
Record Dates: First submitted 2012-01-05; First posted 2012-01-26 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Cervicobrachial Neuralgia; Cervical Discopathy
Keywords: Cervicobrachial; neuralgia; symptomatic cervical discopathy
MeSH Terms: conditions — Brachial Plexus Neuritis; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiculopathy Cervical: Radiculopathy, Cervical
  Interventions: Device: Cervical arthroplasty surgery with Granvia-C

INTERVENTIONS:
Device: Cervical arthroplasty surgery with Granvia-C — Discectomy and Cervical arthroplasty according to standard practice of the surgeon

SUMMARY:
This is a prospective clinical study to assess the performance of the prosthesis according to a composite success criterion. The clinical and functional results and the patient's quality of life up to 24 months of follow-up will also be recorded.

Granvia-c is a device NOT FDA-approved and NOT under investigation in the USA.

DETAILED DESCRIPTION:
Anterior cervical arthrodesis has been widely used to treat the degenerative cervical spine. Although the results of ACDF are generally in the good to excellent range, interbody fusion of the cervical spine after cervical discectomy, aside from causing restriction of neck movements, also accelerates degeneration of adjacent disc levels because of the increased stress from fusion. Long-term radiographic follow-up of patients with anterior cervical fusion has demonstrated degenerative changes in the non-fused segments of the spine including disc space narrowing and osteophyte formation.

To conclude, fusion provokes a functional overload of the discs bordering the fusion that is directly correlated to the number of fused levels. Radiographic observations show a greater mechanical stress on the discs, especially in the arthrodeses involving more than one level.

Artificial discs were designed to replace the entire intervertebral disc and to preserve the physiological motion of the operated level. Several prostheses with different concepts were commercialized. Published clinical studies reported a preserved motion and improved clinical results (Neck Disability Index, Pain Visual Analogic Scale, Quality of Life).

The cervical disc prosthesis GRANVIA®-C was designed to replace the intervertebral discs of the cervical spine, to restore the disc height and to restore segmental motion.

A prospective clinical study has been set up to evaluate the performance of the prosthesis

Granvia-c is a device NOT FDA-approved and NOT under investigation in the USA.

ELIGIBILITY:
Inclusion Criteria:

* Cervicobrachial neuralgia due to symptomatic cervical discopathy
* Presence of pain (arm or arm and neck) and/or a neurologic deficit with a radiographic confirmation (by CT, MRI, X-ray, etc.) of any of the following:

  * Herniated nucleus pulposus
  * Spondylosis (defined by the presence of osteophytes)
* Degenerative Disc Disease at a single level or 2-level(s) adjacent or not between C3 and C7

Exclusion Criteria (non exhaustive):

* Asymptomatic degenerative disc disease (DDD)
* DDD of 3-levels or more
* Axial neck pain as the solitary symptom
* Severe spondylosis at the level to be treated by arthroplasty as
* Characterized by any of the following:

  * Bridging osteophytes
  * A loss of disc height greater than 50% (compared to adjacent levels)
  * Absence of motion (<2°)
* Any prior spine surgery at any cervical level, especially fusion procedure; views) for the level operated by arthroplasty
* Tumor
* Deformity or fracture of the cervical vertebrae
* Active systemic infection or infection at the operative site(s)

  * Pregnant or interested in becoming pregnant in the next three years;
  * Advanced emphysema, Alzheimer's disease or other medical conditions that would interfere with patient self-assessment of function, pain or quality of life

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: People with Cervicobrachial neuralgia due to symptomatic cervical discopathy
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Composite criterion of success | 24Months
  the success is defined by a composite criterion of 4 points. The surgery will be a success only if there is:
  * A 15-point improvement in the NDI score from the preoperative baseline score
  * Maintenance or improvement of the pre-op baseline neurological status
  * Absence of secondary surgical intervention
  * Absence of serious adverse event

SECONDARY OUTCOMES:
Radiologic evaluation of the motion | Preop, 3M, 12M and 24M
  Radiologic evaluation of the motion of the operated level(s) and comparison to the motion of the adjacent levels,
Evaluation of potential peri and post-operative adverse events related or not to prosthesis. | preop, 3M, 12M, 24M
Evaluation of satisfaction | Preop, 3M, 12M and 24M
  Evaluation of satisfaction with Patient Satisfaction Index
Evaluation of the time to return to activities (normal activity, work, sport activity) | preop, 3M, 12M, 24M
Evaluation of Pain | Preop, 3M, 12M and 24M
  Evaluation of pain with Visual Analog Scales
cervical alignment | Preop, 3M, 12M and 24M
  Radiologic evaluation of the global cervical alignment
disc height | Preop, 3M, 12M and 24M
  Radiologic evaluation of the disc height of the operated level(s)
Radiologic adverse events | Preop, 3M, 12M and 24M
  Radiologic evaluation of adverse events such as migration, subsidence

CONTACTS AND LOCATIONS:
Overall Officials: John Yeh, MD, Principal Investigator — Royal London Hospital, UK; Frédéric Schils, MD, Principal Investigator — CHC Liège, Belgium; Hans Meisel, MD, Principal Investigator — Halle Klinike, Germany; Patrick Guérin, MD, Principal Investigator — University Hospital, Bordeaux
Locations (3):
- CHR Namur, Namur, Belgium
- France (2):
  - Tripode Hospital, Bordeaux
  - Clairval hospital, Marseille